CLINICAL TRIAL: NCT02785042
Title: Optical Coherence Tomography (OCT) Reference Data Collection Study (S-2015-3)
Status: Terminated | Type: Observational
Why Stopped: difficulty in recruiting older subjects
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: S-2015-3-hi
Record Dates: First submitted 2016-05-19; First posted 2016-05-27 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2023-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal healthy volunteers: imaging with Heidelberg Spectralis OCT
  Interventions: Device: Heidelberg Spectralis OCT

INTERVENTIONS:
Device: Heidelberg Spectralis OCT — OCT imaging

SUMMARY:
This prospective, single-arm clinical multicenter study intends to measure normal structural parameters of the optic nerve head, the peripapillary retinal nerve fiber layer, and the macula using the Heidelberg Spectralis OCT device. This study is conducted in Hispanic descent volunteers. The main goal of the study is to provide the range of these structural parameters in normal eyes. The study will include at least 240 normal volunteers.

DETAILED DESCRIPTION:
This prospective, single-arm clinical multicenter study intends to measure normal structural parameters of the optic nerve head, the peripapillary retinal nerve fiber layer, and the macula using the Heidelberg Spectralis OCT device. This study is conducted in Hispanic descent volunteers. The main goal of the study is to provide the range of these structural parameters in normal eyes. The study will include at least 240 normal volunteers; up to 10 study sites will recruit subjects. Overall an approximately equal age distribution from 18 to 90 years and an approximately equal number of females and males will be enrolled (approximately 40-60% females in each age group). All subjects will undergo Spectralis OCT imaging, biometric and ophthalmoscopic examination, disc photography and visual field testing in one single visit, if possible. Repeated perimetry or Spectralis scans may be performed at a second visit within 30 days of the initial visit. All examinations performed on the subjects are non-significant risk procedures.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to undergo the test procedures, give consent, and to follow instructions.
* Signed informed consent
* Age ≥18 to 90.
* Healthy eye without prior intraocular surgery (except cataract surgery and Laser in Situ Keratomileusis) and without clinically significant vitreal, retinal or choroidal diseases, clinically significant diabetic retinopathy (subject may have diabetes), or disease of the optic nerve. Small drusen are acceptable in older subjects.
* Hispanic decent (self-reported)
* Negative history of glaucoma (not including family history)
* Intraocular pressure ≤21mmHg.
* Best corrected visual acuity ≥20/40.
* Refraction between +6 and -6 diopters and astigmatism ≤ 2 diopters.
* Axial length ≤ 26.0 mm (by optical biometry)
* Normal visual field with Glaucoma Hemifield Test and Mean Deviation within normal limits or not abnormal visual field by judgment of the ophthalmologist / optometrist
* Clinically normal appearance of the optic disc, with normal appearing neuroretinal rim with respect to color and shape. The optic disc is examined ophthalmoscopically and by evaluation of stereo photographs.
* If both eyes are eligible, both eyes enter the study.

Exclusion Criteria:

* Vulnerable subjects (as defined in ISO 14155 GCP) with the exception of employees of the site, and, if applicable, students of the respective university. Staff that is listed on the delegation form are excluded from participation.
* Subjects unable to read or write
* Unreliable visual field. The reliability indices should be used as guide as well as the perimetrist's notes.
* Unusable disc stereo photos.
* Inability to undergo the tests.
* Insufficient quality of Spectralis OCT images (this is not determined until after Spectralis OCT examination, and is an unusual circumstance).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy eyes without prior intraocular surgery (except cataract surgery and Laser in Situ Keratomileusis) and without clinically significant vitreal, retinal or choroidal diseases, clinically significant diabetic retinopathy (subject may have diabetes), or disease of the optic nerve from subjects of hispanic decent (self-reported).
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-07 (Actual)

PRIMARY OUTCOMES:
Bruch-Membrane-Opening - Minimum Rim Width (µm) | Baseline
  Bruch-Membrane-Opening - Minimum Rim Width (µm)
Bruch-Membrane-Opening - Minimum Rim Area (µm^2) | Baseline
  Bruch-Membrane-Opening - Minimum Rim Area (µm^2)
Peripapillary Retinal Nerve Fibre Layer Thickness (µm) | Baseline
  Peripapillary Retinal Nerve Fibre Layer Thickness (µm)

CONTACTS AND LOCATIONS:
Overall Officials: Balwantray Chauhan, OD, Principal Investigator — Department of Ophthalmology and Visual Sciences Dalhousie University
Locations (8):
- United States (8):
  - University California San Diego, La Jolla, California
  - Assil Eye Institute, Santa Monica, California
  - North Bay Eye Associates, Santa Rosa, California
  - Mid Florida Eye Center Clinic, Mt. Dora, Florida
  - Illinois Eye Institute, Illinois College of Optometry, Chicago, Illinois
  - SUNY College of Optometry, New York, New York
  - Ophthalmic Consultants of Long Island-Valley Stream, Valley Stream, New York
  - Wills Eye Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No